CLINICAL TRIAL: NCT03213080
Title: Discovery of the Impact of Targeted Lung Denervation (TLD) on the Severe and Very Severe COPD Population
Acronym: DISCOVER TLD
Status: Withdrawn | Type: Observational
Why Stopped: Not initiated
Sponsor: Nuvaira, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D0476
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: COPD
Keywords: Targeted Lung Denervation; TLD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TLD Procedure: All subjects who are enrolled and meet the eligibility criteria will undergo Targeted Lung Denervation (TLD). TLD is a bronchoscopically-guided, minimally-invasive procedure using the Nuvaira™ Lung Devervation System. The Nuvaira System is intended for the long-term maintenance treatment of airway obstruction associated with COPD. TLD uses radiofrequency (RF) energy to ablate the airway nerve trunks of the vagus nerves that travel parallel to and outside of the main bronchi and into the lungs. Ablation of the nerves opens the airways and makes breathing easier.
  Interventions: Device: Targeted Lung Denervation (TLD)

INTERVENTIONS:
Device: Targeted Lung Denervation (TLD) — Targeted Lung Denervation (TLD) procedure.

SUMMARY:
The DISCOVER TLD study is a multicenter, prospective, single-arm study designed to record the clinical outcomes of the CE-marked Nuvaira™ Lung Denervation System, in a subset of its CE-marked approved indication. This study is being conducted in Europe.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the overall COPD patient experience with the Nuvaira™ Lung Denervation System and allow for the continued collection of safety and effectiveness data on the CE-marked product. The study is a multicenter, prospective, single-arm study designed to include patients, on average, who fall within a more severe stage of COPD, defined as 20-45% FEV1 percent predicted. Subjects will remain on respiratory medications per their standard of care and will be followed and tested per standard of care throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD with 20% ≤ FEV1 ≤ 45% and FEV1/FVC < 70% (post-bronchodilator)
* History of long-term smoking, but non-smoking for a minimum of 2 months prior to study consent
* Patient is a candidate for bronchoscopy
* Patient agrees to all follow-up and provides written informed consent.

Exclusion Criteria:

* Presence of lung or chest implants (eg. metal stent, valves, coils)
* Pregnancy
* Pre-existing pulmonary hypertension
* Patient has a pacemaker, internal defibrillator, or other implantable electronic device
* Inappropriate bronchial anatomy for procedure (per CT scan)
* Previous abdominal surgical procedures on stomach, esophagus or pancreas
* Previous treatment with TLD Therapy (in same areas)
* Known allergy to bronchoscopy or general anesthesia medications
* Inability to tolerate single lung ventilation for at least 2 min, 30 sec
* Patient has a GCSI score of ≥ 18 at time of screening visit

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of advanced COPD [20% ≤ FEV1 ≤ 45% and FEV1/FVC < 70% (post-bronchodilator)] who are no longer smoking (quit at least 2 months prior to registry consent) and are able to undergo general anesthesia. All subjects will undergo a CT scan to determine whether bronchial anatomy is appropriate for TLD procedure.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life (QOL) | 6 months; 12 months; 24 months post-procedure
  Changes in the St. George's Respiratory Questionnaire for COPD patients (SGRQ-C) over time will be assessed. Comparisons will be made to baseline score.

SECONDARY OUTCOMES:
Changes in Pulmonary Function | 6 months, 12 months, 24 months post-procedure
  Basic spirometry tests including FEV1, FVC, forced impulse oscillometry, nitrogen wash-out measures will be performed per standard of care over time. Comparisons will be made to baseline measures.
Change in 6-Minute Walk Test | 6 months, 1 year, 2 years
  Change in 6MWT over time
Respiratory-related Adverse Events | 24 months
  Respiratory-related adverse events will be collected throughout the registry. Rates of respiratory-related adverse events will be reported and compared to historical data.
Freedom from Device-related Adverse Events | Peri-procedure (within 7 days); 1 month and 6 months
  Device-related adverse events will be collected through 6 months post-procedure. The number of subjects free from a device-related adverse event will be reported.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Nuvaira Website with description of TLD procedure — https://www.nuvaira.com/